CLINICAL TRIAL: NCT02586740
Title: Retrospective Review of Anesthetic Considerations for Pulmonary Artery Rehabilitation
Status: Completed | Type: Observational
Sponsor: Aymen N Naguib (Other)
Responsible Party: Sponsor-Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB15-00914
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Pulmonary Artery Stenosis; Tetralogy of Fallot; Pulmonary Atresia
MeSH Terms: conditions — Stenosis, Pulmonary Artery; Tetralogy of Fallot; Pulmonary Atresia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pulmonary artery rehabilitation: Patients with pulmonary artery stenosis or small pulmonary arteries following surgical repair for tetralogy of Fallot with pulmonary atresia and major aortopulmonary collaterals undergoing cardiac catheterization.
  Interventions: Procedure: Pulmonary artery rehabilitation

INTERVENTIONS:
Procedure: Pulmonary artery rehabilitation

SUMMARY:
Pulmonary artery rehabilitation procedure is done frequently in the catheterization suite for patients with pulmonary artery stenosis or small pulmonary arteries following surgical repair for patients with tetralogy of Fallot with pulmonary atresia and major aortopulmonary collaterals. Considering that the investigators' institution is a major center for treating these cases, the investigators wanted to do a retrospective review of the investigators' data to share the investigators' anesthetic management of these procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent pulmonary artery angioplasty during the period between October 1st 2010 and October 1st 2015 at NCH.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pulmonary artery stenosis or small pulmonary arteries following surgical repair for tetralogy of Fallot with pulmonary atresia and major aortopulmonary collaterals.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience hemorrhage | During catheterization procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States